CLINICAL TRIAL: NCT02949089
Title: An Open Label, Dose Escalation Study of ACH04 to Assess the Safety and Tolerability in Healthy Adults Subjects
Brief Title: ACH04 to Assess the Safety and Tolerability in Healthy Adults Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACH-PSD-01(04/11)
Record Dates: First submitted 2011-05-03; First posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Diarrhea
Keywords: safety; tolerability; rising multiple doses; ACH04; adult; male
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACH04 (Experimental): Dosage: 1 capsule, PO, 24/24h for 10 days.
  Interventions: Drug: ACH04

INTERVENTIONS:
Drug: ACH04 — The subjects will receive the study medication in each group

SUMMARY:
This study intends to provide information on the safety and tolerability of repeated oral doses of ACH04. A phase I, single-center, first in human, open-label, dose escalation study of ACH04 to assess the safety and tolerability in healthy adults subjects is selected to best address the study goals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be healthy males subjects between 18 and 50 years of age;
* Subjects must be in good healthy as determined by a medical history, physical examination and clinical laboratory evaluations;
* Subjects will, prior to any study related activities, have given their written informed consent to participate in the study and to abide by the stdy restrictions.

Exclusion Criteria:

* Subjects with hypersensitivity known to Psidium guajava L. or history of serious adverse events;
* Subjects who have a significant history of alcoholism or drug/chemical abuse;
* Subjects who have body mass index < 18 or > 30;
* Subjects who have received any medications that is known to have a toxic potential well defined in large organs within the past 3 months prior the study start;
* Subjets who doesn´t agree to use, for the duration of the study, a barrier contraceptive;
* Subjects who were hospitalized for any reason in the six week prior the study start;
* Subjects who, in the opinion of the investigator, should not participate in the study, including subjects suspected for whatever reason of not being able to comply with the requirements of the protocol;
* Subjects who are participating in a clinical trial or have participated in a clinical study involving administration of an investigational drug, within one year;
* Subjects who are relatives of employees from the sponsor and the site, respectively;
* Subjects with, or with a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological, dermatological or other major disorders as determined by the Investigator;
* Any finding of clinical observation (anamnesis and physical evaluation), laboratory abnormality, who in the investigator opinion, may jeopardize the subjects or interfere with the study goals.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of rising multiple doses of ACH04 | up to 39 days
  Evaluate the occurrence of adverse events, Assess safety through laboratory tests and Assess safety through electrocardiogram

CONTACTS AND LOCATIONS:
Locations (1):
- UNIFAC, Fortaleza, Ceará, Brazil